CLINICAL TRIAL: NCT02647268
Title: Effect of Magnesium Sulphate Pre-exposure on Oxytocin-induced Contractility in Desensitized Human Myometrium - an in Vitro Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-01
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Oxytocin; Magnesium sulphate
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (no oxytocin) pretreatment (No Intervention): The myometrial samples are bathed in physiological saline solution (PSS).
- Magnesium Sulphate (Active Comparator): The myometrial samples are bathed in a 3.5mM magnesium sulphate solution.
  Interventions: Drug: Magnesium Sulphate
- Magnesium Sulphate + oxytocin (Active Comparator): The myometrial samples are bathed in a 3.5mM magnesium sulphate plus 10-5M oxytocin solution.
  Interventions: Drug: Oxytocin; Drug: Magnesium Sulphate

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 10-5M solution
  Other Names: pitocin
  Arms: Magnesium Sulphate + oxytocin
Drug: Magnesium Sulphate — Magnesium sulphate, 3.5mM solution
  Arms: Magnesium Sulphate; Magnesium Sulphate + oxytocin

SUMMARY:
Postpartum hemorrhage (PPH) is the loss of more than 500ml of blood within 24 hours after delivery. It is a major cause of maternal morbidity and mortality across the globe.

Oxytocin is a naturally-occurring hormone that causes the uterus to contract, thereby causing labor. A synthetic form of oxytocin is used in obstetric medicine in the same way. It causes the uterus to contract by acting at the oxytocin receptor (OTR). It is used for both the prevention and the treatment of PPH. By causing the uterus to contract, it constricts the blood vessels within it, thus reducing bleeding.

Oxytocin is also used to augment labor in women with slow labor progression. Desensitization of the OTR after prolonged exposure to oxytocin occurs, leading to reduced contractions of the uterus with the same doses of oxytocin. This has been demonstrated in previous studies done by the investigators. The resultant need for a higher oxytocin dose to cause adequate uterine contraction has also been demonstrated in laboring women having received oxytocin for labor augmentation.

Magnesium sulphate (MgSO4) is widely used within obstetric medicine. It is used for seizure prevention and treatment in preeclampsia and eclampsia, and is used for fetal neuroprotection in preterm labor, to reduce the risk of cerebral palsy. It is well-known to have a relaxant effect on uterine muscle, and as such, has been used as a tocolytic agent in preterm labour to prevent premature contractions and premature delivery. The effect of MgSO4 on contractions in oxytocin pre-treated myometrium has not been fully elucidated with human lab studies. There are suggestions it may lead to increased oxytocin requirements or increased postpartum hemorrhage (PPH) in preeclamptic patients. This bears significance in the preeclamptic and eclamptic populations who are likely to be receiving MgSO4 in combination with oxytocin.

The investigators hypothesize that MgSO4 will reduce uterine contractions in oxytocin pre-treated myometrium, as well as untreated myometrium, and higher oxytocin doses will be needed to produce equivalent contractions. This will help us to better understand the implications of the use of these drugs together in the clinical setting.

DETAILED DESCRIPTION:
MgSO4 is known to cause relaxation of uterine muscle in the doses used for preeclampsia and eclampsia and fetal neuroprotection. In these clinical settings, after delivery, oxytocin is often given to prevent or treat PPH. There is evidence that patients with preeclampsia already have a higher risk of PPH than non-preeclamptic patients. In the presence of the effects of MgSO4 treatment on the uterus, PPH could be worse in theory. If patients have had oxytocin-augmented labor, then the desensitization effect on the uterus also comes into play. Performing this study in vitro will allow us to assess the effects on the uterine muscle of MgSO4 in oxytocin-desensitized tissue samples.

Scientific evidence on pregnancy outcomes in these patients is timely and important. A study of myometrial contractility under controlled conditions is likely to provide us with information on the interactions between oxytocin and MgSO4 that occurs in many clinical scenarios, eliminating any confounders that could be encountered in clinical settings. The investigators hope to determine the myometrial contraction patterns induced by oxytocin in the presence of MgSO4, including in myometrial specimens pre-treated with oxytocin plus MgSO4, to mimic the clinical scenarios in preeclampsia and fetal neuroprotection. This will expand the depth of our understanding of the desensitization phenomenon, and could provide valuable insight into the mechanism responsible for PPH in these patient populations. This study will form a basis for future modifications in oxytocin augmentation regimens and pharmacotherapy for control of uterine atony and PPH in these patient populations being simultaneously treated with MgSO4.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary Cesarean delivery or first repeat Cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients who had previous uterine surgery or more than one previous Cesarean delivery
* Patients with any condition predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, bleeding diathesis, chorioamnionitis, or a previous history of postpartum bleeding
* Emergency Cesarean section in labor
* Patients with medical/pregnancy related conditions, such as diabetes, preeclampsia and essential hypertension

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Motility Index | 2 hours
  Motility index (MI) takes into account both the amplitude and frequency of the myometrial contraction. It is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 2 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 2 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Onwochei DN, Carvalho JCA, Luca A, Kingdom J, Balki M. Effect of magnesium sulfate on oxytocin-induced contractility in human myometrium: an in vitro study. Can J Anaesth. 2017 Jul;64(7):744-753. doi: 10.1007/s12630-017-0867-3. Epub 2017 Mar 30. PMID 28361390